CLINICAL TRIAL: NCT03286777
Title: Increasing the Oral Bioavailability of 6-prenylnaringenin by Micellar Solubilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS-PF2-2017
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Safety of Native vs. Micellar 6-PN After Oral Intake; Pharmacokinetics of Native vs. Micellar 6-PN After Oral Intake; PBMC Activity After Native vs. Micellar 6-PN Oral Intake
Keywords: 6-prenylnaringenin; Bioavailability; Pharmacokinetics; PBMC

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Mannitol and silicon dioxide
  Interventions: Dietary Supplement: Placebo
- Native 6-prenylnaringenin (Experimental): 250 mg native 6-PN plus mannitol and silicon dioxide
  Interventions: Dietary Supplement: Native 6-prenylnaringenin
- Micellar 6-prenylnaringenin (Experimental): 250 mg 6-PN in a micellar formulation with Tween-80 as adjuvant
  Interventions: Dietary Supplement: Micellar 6-prenylnaringenin

INTERVENTIONS:
Dietary Supplement: Placebo — Mannitol and silicon dioxide capsules
  Arms: Placebo
Dietary Supplement: Native 6-prenylnaringenin — 250 mg native 6-PN plus mannitol and silicon dioxide capsules
  Arms: Native 6-prenylnaringenin
Dietary Supplement: Micellar 6-prenylnaringenin — 250 mg 6-PN in a micellar formulation with Tween-80 as adjuvant capsules
  Arms: Micellar 6-prenylnaringenin

SUMMARY:
Micellar encapsulation will be tested to increase the oral bioavailability in humans of 6-prenylnaringenin (6-PN) from hops (Humulus lupulus). The study follows a single dose (250 mg 6-PN), placebo controlled, randomized, double-blind, three armed crossover study design with ≥2-week washout periods. Plasma, urine and PBMC samples will be collected at intervals up to 24 h after intake of the native compound, the micellar formulation or placebo. The safety, pharmacokinetics and impact of oral prenylflavonoids on PBMC survival will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with blood chemistry values within normal ranges
* Age: 18-45 years
* BMI: 19-25 kg/m2

Exclusion Criteria:

* Pregnancy or lactation
* Alcohol and/or drug abuse
* Use of dietary supplements or any medications, except contraceptives
* Any known malignant, metabolic and endocrine diseases
* Previous cardiac infarction
* Dementia
* Participation in a clinical trial within the past 6 weeks prior to recruitment
* Physical activity of more than 5 h/wk

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Mean area under the curve (AUC) of plasma concentration vs. time of total 6-PN [nmol/L*h] | 0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 24 h post dose
  Total 6-PN determined after deconjugation with beta-glucuronidase/sulphatase
Mean maximum plasma concentration (Cmax) of total 6-PN [nmol/L] | 0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 24 h post dose
  Total 6-PN determined after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total 6-PN [h] | 0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 24 h post dose
  Total 6-PN determined after deconjugation with beta-glucuronidase/sulphatase
Cumulative urinary excretion of total 6-PN [nmol/g creatinine] | 0 h - 24 h post dose
  Total 6-PN determined after deconjugation with beta-glucuronidase/sulphatase
Cell count (dead cells/ml and living cells/ml) of PBMCs after 6-PN administration | 0 h, 6 h, and 24 h post dose
Cell viability of PBMCs after 6-PN administration | 0 h, 6 h, and 24 h post dose

SECONDARY OUTCOMES:
Serum aspartate transaminase activity [U/L] | 0 h, 4 h, 24h post-dose
Serum alanine transaminase activity [U/L] | 0 h, 4 h, 24h post-dose
Serum gamma-glutamyl transferase activity [U/L] | 0 h, 4 h, 24h post-dose
Serum alkaline phosphatase activity [U/L] | 0 h, 4 h, 24h post-dose
Serum bilirubin | 0 h, 4 h, 24h post-dose
Serum uric acid [mg/dL] | 0 h, 4 h, 24h post-dose
Serum creatinine [mg/dL] | 0 h, 4 h, 24h post-dose
Serum total cholesterol [mg/dL] | 0 h, 4 h, 24h post-dose
Serum HDL cholesterol [mg/dL] | 0 h, 4 h, 24h post-dose
Serum LDL cholesterol [mg/dL] | 0 h, 4 h, 24h post-dose
Serum triacylglycerols [mg/dL] | 0 h, 4 h, 24h post-dose
LDL/HDL cholesterol ratio | 0 h, 4 h, 24h post-dose
Glomerular filtration rate [mL/min] | 0 h, 4 h, 24h post-dose
Serum glucose [mg/dL] | 0 h, 4 h, 24h post-dose
Hemoglobin [g/dL] | 0 h, 24 h post-dose
Mean corpuscular hemoglobin concentration [g/dL] | 0 h, 24 h post-dose
Mean corpuscular hemoglobin [pg] | 0 h, 24 h post-dose
Mean corpuscular volume [fL] | 0 h, 24 h post-dose
Hematocrit [%] | 0 h, 24 h post-dose
Erythrocytes [/pL] | 0 h, 24 h post-dose
Thrombocytes [/nL] | 0 h, 24 h post-dose
Leucocytes [/nL] | 0 h, 24 h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frank, Prof. Dr., Principal Investigator — University of Hohenheim; Sascha Venturelli, Dr. med. Dr. rer. nat., Principal Investigator — University Hospital, Eberhard Karls University Tuebingen, Germany; Christian Busch, Dr. med., Principal Investigator — University Hospital, Eberhard Karls University Tuebingen, Germany
Locations (2):
- Germany (2):
  - University of Hohenheim, Stuttgart, Baden-Wurttemberg
  - Eberhard Karls University Tuebingen, Tübingen, Baden-Wurttemberg

REFERENCES:
- See also: Website of the research group — http://www.nutrition-research.de/